CLINICAL TRIAL: NCT02666352
Title: A Two-Part, Open-Label Study to Investigate the Single-Dose Pharmacokinetics of MK-3682 and MK-8408 When Coadministered to Subjects With Moderate and Severe Hepatic Insufficiency
Brief Title: A Study of the Pharmacokinetics of Uprifosbuvir (MK-3682) and Ruzasvir (MK-8408) in Participants With Moderate and Severe Hepatic Insufficiency (MK-3682-029)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-029
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — uprifosbuvir; ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate HI Participants (Experimental): On Day 1, participants with moderate HI will receive a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir
- Severe HI Participants (Experimental): On Day 1, participants with severe HI will receive a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir
- Healthy Participants (Experimental): On Day 1, participants with normal hepatic function will receive a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
  Interventions: Drug: Uprifosbuvir; Drug: Ruzasvir

INTERVENTIONS:
Drug: Uprifosbuvir — A single dose of uprifosbuvir 450 mg (given as three 150-mg tablets) taken by mouth.
  Other Names: MK-3682
Drug: Ruzasvir — A single dose of ruzasvir 60 mg (given as six 10-mg capsules) taken by mouth.
  Other Names: MK-8408

SUMMARY:
This is a non-randomized, open-label, single-dose study to evaluate the pharmacokinetics (PK) of uprifosbuvir (MK-3682), the M5 and M6 metabolites of uprifosbuvir, and ruzasvir (MK-8408), in participants with moderate hepatic insufficiency (HI), participants with severe HI, and age-matched healthy control participants.

ELIGIBILITY:
Inclusion Criteria:

HI Participants Only:

* Has a diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) HI features of cirrhosis;
* Part 1 only: Participant's score on the Child-Pugh scale ranges from 7 to 9 (moderate HI) at study start.
* Part 2 only: Participant's score on the Child-Pugh scale ranges from 10 to 15 (severe HI) at study start.

All Participants:

* Body mass index (BMI) ≥19 and ≤ 40 kg/m^2;
* Continuous non-smokers or moderate smokers (of fewer than 20 cigarettes/day or the equivalent). Participants must agree to consume no more than 10 cigarettes or equivalent/day from the time of screening and throughout the period of sample collection;
* Health is judged to be stable based on medical history (except for the hepatic impairment condition), physical examination, vital signs, electrocardiogram (ECGs), and laboratory safety tests;
* For female participants of childbearing potential: either sexually inactive for 14 days prior to study start and throughout study or be using an acceptable birth control method;
* Female participants who are sexually inactive, but become sexually active during the course of the study must agree to use a double physical barrier method (e.g., condom and diaphragm) and a chemical barrier (e.g., spermicide) from the time of the start of sexual activity through completion of the study;
* Vasectomized or non-vasectomized male participants must agree to use a condom with spermicide or abstain from sexual intercourse from dosing until 90 days after dosing;
* Male participants must agree not to donate sperm from dosing until 90 days after dosing;
* Able to swallow multiple tablets and capsules.

Exclusion Criteria:

HI Participants Only:

* Presence of moderate or severe renal insufficiency (estimated glomerular filtration rate [eGFR] ≤50 mL/min/1.73 m^2 calculated according to the Modification of Diet in Renal Disease [MDRD] study equation);
* Presence of drug abuse within the past 6 months prior to dosing.

Healthy Participants Only:

* Presence of moderate or severe renal insufficiency (eGFR ≤60 mL/min/1.73 m^2 calculated according to the MDRD study equation);
* History or presence of alcoholism or drug abuse within the past 2 years prior to dosing;

All Participants:

* Is mentally or legally incapacitated or has significant emotional problems at the time of study start or expected during the study;
* History or presence of clinically significant medical or psychiatric condition or disease;
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds;
* Female participants who are pregnant or lactating;
* Positive results at study start for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
* Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) for the prohibited time period;
* Has taken amiodarone at any time in their life;
* Donation of blood >500 mL or had significant blood loss within 56 days prior to the dose of study drugs;
* Plasma donation within 7 days prior to the dose of study drugs;
* Dosed in another clinical trial within 28 days prior to dosing of study drugs;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderate hepatic insufficiency (HI), severe HI, and healthy controls were recruited at 2 study centers in the United States.
Groups:
- Moderate HI Participants: Participants with moderate HI (Child-Pugh score 7 to 9) received a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
- Severe HI Participants: Participants with severe HI (Child-Pugh score 10 to 15) received a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
- Healthy Participants: Participants with normal hepatic function received a single oral dose of 450 mg uprifosbuvir (3 x 150 mg tablets) and 60 mg ruzasvir (6 x 10 mg capsules) following an overnight fast.
Period: Overall Study
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (8.7) | 55.4 (8.2) | 57.6 (6.3) | 57.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 6 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Drug Plasma Concentration-Time Curve From Start of Dosing to Time of the Last Quantifiable Sample (AUC0-last) of Uprifosbuvir
Description: AUC0-last is a measure of the mean plasma drug concentration from time of dosing to the last quantifiable sample. The AUC0-last for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 5.34 [3.55 to 8.05] | 8.02 [5.32 to 12.1] | 3.74 [2.48 to 5.63]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.43, 90% CI 2-sided [0.89 to 2.31]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 2.15, 90% CI 2-sided [1.33 to 3.47]

2. Primary Outcome: Area Under the Drug Plasma Concentration-Time Curve From Start of Dosing to Infinity (AUC0-inf) of Uprifosbuvir
Description: AUC0-inf is a measure of the mean plasma drug concentration from time of dosing to infinity. The AUC0-inf for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 5.39 [3.57 to 8.12] | 8.09 [5.37 to 12.2] | 3.76 [2.50 to 5.68]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.43, 90% CI 2-sided [0.88 to 2.31]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 2.15, 90% CI [1.33 to 3.48]

3. Primary Outcome: Area Under the Plasma Drug Concentration-Time Curve From Start of Dosing to 24 Hours Post-Dose (AUC0-24hr) of Uprifosbuvir
Description: AUC0-24hr is a measure of the mean plasma drug concentration from time of dosing to 24 hours post-dose. The AUC0-24hr for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 5.35 [3.55 to 8.05] | 8.02 [5.33 to 12.1] | 3.74 [2.48 to 5.63]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.43, 90% CI 2-sided [0.89 to 2.31]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 2.15, 90% CI 2-sided [1.33 to 3.47]

4. Primary Outcome: Maximum Plasma Drug Concentration (Cmax) of Uprifosbuvir
Description: Cmax is the maximum observed plasma drug concentration after dosing. The Cmax for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 1560 [1030 to 2360] | 2130 [1410 to 3240] | 1180 [778 to 1790]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.32, 90% CI 2-sided [0.81 to 2.15]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.81, 90% CI 2-sided [1.11 to 2.94]

5. Primary Outcome: Plasma Drug Concentration at 24 Hours (C24hr) of Uprifosbuvir
Description: C24hr is a measure of plasma drug concentration 24 hours after dosing. The C24hr of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 7.01 [0.00 to 26.9] | 8.56 [0.00 to 85.5] | 2.55 [0.00 to 22.3]

6. Primary Outcome: Time to Reach Cmax (Tmax) of Uprifosbuvir
Description: Tmax is the time required to reach maximum plasma drug concentration (i.e., Cmax). The Tmax for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 1.00 [0.50 to 4.00] | 0.50 [0.50 to 1.50] | 1.25 [0.50 to 3.00]

7. Primary Outcome: Apparent Terminal Half-Life (t1/2) of Uprifosbuvir
Description: t1/2 is a measure of how long it takes to clear 50% of drug after reaching Cmax. The t1/2 for uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 3.66 (21.7) | 3.56 (47.5) | 3.17 (38.5)

8. Primary Outcome: Apparent Total Clearance From Plasma After Oral Administration (CL/F) of Uprifosbuvir
Description: CL/F is a measure of the apparent rate at which drug is removed from the body via renal, hepatic, and other clearance pathways after oral administration. The CL/F of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
L/hr | 153 (39.9) | 102 (61.1) | 219 (77.6)

9. Primary Outcome: Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) of Uprifosbuvir
Description: Vz/F is the apparent volume of distribution during the terminal phase after non-intravenous administration. The Vz/F of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
L | 809 (43.8) | 524 (57.0) | 1000 (83.0)

10. Primary Outcome: AUC0-last of Uprifosbuvir Metabolite M5
Description: AUC0-last is a measure of the mean plasma drug concentration from time of dosing to the last quantifiable sample. The AUC0-last for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 6.46 [4.90 to 8.52] | 6.79 [5.15 to 8.95] | 8.11 [6.15 to 10.7]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.80, 90% CI 2-sided [0.58 to 1.10]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.84, 90% CI 2-sided [0.61 to 1.16]

11. Primary Outcome: AUC0-inf of Uprifosbuvir Metabolite M5
Description: AUC0-inf is a measure of the mean plasma drug concentration from time of dosing to infinity. The AUC0-inf for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 6.78 [5.15 to 8.93] | 7.22 [5.48 to 9.50] | 8.44 [6.41 to 11.1]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.80, 90% CI 2-sided [0.58 to 1.11]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.86, 90% CI [0.62 to 1.18]

12. Primary Outcome: AUC0-24hr of Uprifosbuvir Metabolite M5
Description: AUC0-24hr is a measure of the mean plasma drug concentration from time of dosing to 24 hours post-dose. The AUC0-24hr for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 2.41 [1.85 to 3.13] | 2.28 [1.75 to 2.96] | 3.12 [2.40 to 4.05]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.77, 90% CI 2-sided [0.57 to 1.05]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.73, 90% CI 2-sided [0.54 to 0.99]

13. Primary Outcome: Cmax of Uprifosbuvir Metabolite M5
Description: Cmax is the maximum observed plasma drug concentration after dosing. The Cmax for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 169 [130 to 220] | 151 [117 to 197] | 203 [156 to 264]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.83, 90% CI 2-sided [0.61 to 1.13]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.75, 90% CI 2-sided [0.55 to 1.01]

14. Primary Outcome: C24hr of Uprifosbuvir Metabolite M5
Description: C24hr is a measure of plasma drug concentration 24 hours after dosing. The C24hr of the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 124 [93.9 to 164] | 122 [92.8 to 162] | 150 [114 to 198]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.83, 90% CI 2-sided [0.60 to 1.15]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.82, 90% CI 2-sided [0.59 to 1.13]

15. Primary Outcome: Lag Time (Tlag) for Uprifosbuvir Metabolite M5
Description: Tlag is a measure of the time delay between drug administration and the onset of absorption, where onset of absorption is defined as "the time point prior to the first observed/measured non-zero plasma concentration". The Tlag of the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm (in this study Tlag was only calculated for the M5 uprifosbuvir metabolite).
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 3.00 [2.00 to 3.00] | 2.53 [2.00 to 3.00] | 2.00 [1.50 to 3.02]

16. Primary Outcome: Tmax of Uprifosbuvir Metabolite M5
Description: Tmax is the time required to reach maximum plasma drug concentration (i.e., Cmax). The Tmax for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 14.00 [12.00 to 18.00] | 16.00 [12.00 to 20.00] | 15.00 [10.00 to 16.00]

17. Primary Outcome: Apparent t1/2 of Uprifosbuvir Metabolite M5
Description: Apparent t1/2 is a measure of how long it takes to clear 50% of drug after reaching Cmax. The t1/2 for the M5 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 24.09 (17.2) | 25.64 (19.2) | 23.59 (9.7)

18. Primary Outcome: AUC0-last of Uprifosbuvir Metabolite M6
Description: AUC0-last is a measure of the mean plasma drug concentration from time of dosing to the last quantifiable sample. The AUC0-last for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 28.6 [22.6 to 36.1] | 27.4 [21.6 to 34.6] | 41.8 [33.0 to 52.9]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.68, 90% CI 2-sided [0.52 to 0.90]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.66, 90% CI 2-sided [0.50 to 0.86]

19. Primary Outcome: AUC0-inf of Uprifosbuvir Metabolite M6
Description: AUC0-inf is a measure of the mean plasma drug concentration from time of dosing to infinity. The AUC0-inf for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 30.1 [23.5 to 38.6] | 28.7 [22.4 to 36.7] | 47.0 [36.7 to 60.2]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.64, 90% CI 2-sided [0.48 to 0.86]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.61, 90% CI [0.46 to 0.82]

20. Primary Outcome: AUC0-24hr of Uprifosbuvir Metabolite M6
Description: AUC0-24hr is a measure of the mean plasma drug concentration from time of dosing to 24 hours post-dose. The AUC0-24hr for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 13.1 [10.6 to 16.1] | 13.2 [10.8 to 16.3] | 16.6 [13.5 to 20.4]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.79, 90% CI 2-sided [0.62 to 1.01]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.80, 90% CI 2-sided [0.63 to 1.02]

21. Primary Outcome: Cmax of Uprifosbuvir Metabolite M6
Description: Cmax is the maximum observed plasma drug concentration after dosing. The Cmax for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 851 [675 to 1070] | 834 [662 to 1050] | 1070 [846 to 1340]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.80, 90% CI 2-sided [0.61 to 1.05]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.78, 90% CI 2-sided [0.60 to 1.03]

22. Primary Outcome: C24hr of Uprifosbuvir Metabolite M6
Description: C24hr is a measure of plasma drug concentration 24 hours after dosing. The C24hr of the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 402 [332 to 487] | 410 [339 to 497] | 564 [465 to 683]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.71, 90% CI 2-sided [0.57 to 0.89]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.73, 90% CI 2-sided [0.58 to 0.91]

23. Primary Outcome: Tmax of Uprifosbuvir Metabolite M6
Description: Tmax is the time required to reach maximum plasma drug concentration (i.e., Cmax). The Tmax for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 6.00 [2.00 to 12.00] | 4.00 [3.00 to 8.00] | 4.00 [3.00 to 6.00]

24. Primary Outcome: Apparent t1/2 of Uprifosbuvir Metabolite M6
Description: Apparent t1/2 is a measure of how long it takes to clear 50% of drug after reaching Cmax. The t1/2 for the M6 metabolite of uprifosbuvir 450 mg (given in combination with ruzasvir 60 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 26.96 (19.4) | 26.45 (31.3) | 33.98 (37.7)

25. Primary Outcome: AUC0-last of Ruzasvir
Description: AUC0-last is a measure of the mean plasma drug concentration from time of dosing to the last quantifiable sample. The AUC0-last for ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 2.30 [1.75 to 3.02] | 2.70 [2.07 to 3.51] | 1.98 [1.52 to 2.58]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio (GMR) = 1.16, 90% CI 2-sided [0.85 to 1.58]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.36, 90% CI 2-sided [1.00 to 1.85]

26. Primary Outcome: AUC0-inf of Ruzasvir
Description: AUC0-inf is a measure of the mean plasma drug concentration from time of dosing to infinity. The AUC0-inf for ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 2.60 [1.99 to 3.41] | 3.32 [2.56 to 4.31] | 2.10 [1.62 to 2.73]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.24, 90% CI 2-sided [0.91 to 1.68]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.58, 90% CI [1.17 to 2.14]

27. Primary Outcome: AUC0-24hr of Ruzasvir
Description: AUC0-24hr is a measure of the mean plasma drug concentration from time of dosing to 24 hours post-dose. The AUC0-24hr for ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
µM*hr | 1.04 [0.729 to 1.49] | 1.05 [0.744 to 1.48] | 1.17 [0.830 to 1.65]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.89, 90% CI 2-sided [0.60 to 1.33]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.90, 90% CI 2-sided [0.60 to 1.34]

28. Primary Outcome: Maximum Plasma Drug Concentration (Cmax) of Ruzasvir
Description: Cmax is the maximum observed plasma drug concentration after dosing. The Cmax for ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 105 [65.6 to 167] | 92.5 [58.9 to 145] | 137 [87.0 to 215]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.77, 90% CI 2-sided [0.45 to 1.30]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 0.68, 90% CI 2-sided [0.40 to 1.14]

29. Primary Outcome: C24hr of Ruzasvir
Description: C24hr is a measure of plasma drug concentration 24 hours after dosing. The C24hr of ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: 24 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
nM | 27.6 [21.4 to 35.7] | 32.4 [25.2 to 41.5] | 23.0 [18.0 to 29.5]
Statistical Analysis 1: Comparison: Moderate HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.20, 90% CI 2-sided [0.90 to 1.60]
Statistical Analysis 2: Comparison: Severe HI Participants vs Healthy Participants; Test type: Other; Geometric least-squares mean ratio = 1.41, 90% CI 2-sided [1.06 to 1.87]

30. Primary Outcome: Tmax of Ruzasvir
Description: Tmax is the time required to reach maximum plasma drug concentration (i.e., Cmax). The Tmax of ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0), and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 3.00 [1.50 to 24.00] | 2.03 [1.50 to 4.00] | 3.00 [2.00 to 4.00]

31. Primary Outcome: Apparent t1/2 of Ruzasvir
Description: Apparent t1/2 is a measure of how long it takes to clear 50% of drug after reaching Cmax. The t1/2 for ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
hr | 38.08 (23.1) | 47.26 (36.6) | 30.43 (14.6)

32. Primary Outcome: CL/F of Ruzasvir
Description: CL/F is a measure of the apparent rate at which drug is removed from the body via renal, hepatic, and other clearance pathways after oral administration. The CL/F of ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
L/hr | 28.4 (36.7) | 20.6 (52.8) | 32.6 (54.6)

33. Primary Outcome: Vz/F of Ruzasvir
Description: Vz/F is the apparent volume of distribution during the terminal phase after non-intravenous administration. The Vz/F of ruzasvir 60 mg (given in combination with uprifosbuvir 450 mg) was calculated for each arm.
Time Frame: Pre-dose (0) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 14, 16, 18, 20, 24, 48, 72, 96, and 120 hours post-dose
Population: All participants are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
Number analyzed (Participants) | 8 | 8 | 8
L | 1560 (49.8) | 1400 (37.9) | 1430 (48.1)

ADVERSE EVENTS:
Time Frame: Up to 14 days
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All participants are included in the safety analysis.
Arm/Group | Moderate HI Participants | Severe HI Participants | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate HI Participants (N=8) | Severe HI Participants (N=8) | Healthy Participants (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will provide separate guidance on the criteria for publication of clinical trial data when contacted for permission to publish.